CLINICAL TRIAL: NCT04121663
Title: Non-inferiority Evaluation of Multicenter, Randomized, Single-blind, Parallel-controlled Clinical Trials on the Safety and Efficacy of Full-suture Anchors for Rotator Cuff Injury and/or Shoulder Instability Surgery
Acronym: MST-002
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-159
Record Dates: First submitted 2019-09-25; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-06

CONDITIONS: Shoulder Instability Rotator Cuff Injury
Keywords: Shoulder instability; Rotator cuff injury
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full seam anchor (Experimental)
  Interventions: Device: Total arthroscopic rotator cuff repair
- Polyether ether ketone bone anchor (Active Comparator)
  Interventions: Device: Total arthroscopic rotator cuff repair

INTERVENTIONS:
Device: Total arthroscopic rotator cuff repair — The equivalence of the two devices was compared by using control and experimental instruments during the operation

SUMMARY:
Multicenter, randomized, single-blind, parallel-controlled non-inferiority assessment for safety and efficacy of rotator cuff injury and/or shoulder instability surgery

DETAILED DESCRIPTION:
This clinical trial compares the clinical effects of rotator cuff injury and/or shoulder instability surgery with the full suture anchor made by Hangzhou Ruijian Mastine Medical Equipment Co., Ltd. and the polyether ether ketone bone anchor system made by Arthrex, Inc., USA, and evaluates the safety and effectiveness of the experimental device in clinical application

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patients ranged from 18 to 75 years (including 18 and 75 years), with no gender limitation
2. Patients with rotator cuff injury and/or instability of the shoulder joint are eligible for surgical indications of suture anchor
3. Subjects were willing and able to sign informed consent

Exclusion Criteria:

1. Patients with severe osteoporosis；
2. A variety of conditions, such as previous infection, suspected infection, current infection, that may or may lead to insufficient implant support or impaired rehabilitation；
3. Those with severe allergic constitution (e.g. severe allergic purpura, asthma, rhinitis, shock, etc.)；
4. Patients with abnormal liver and kidney function [SGPT (ALT) or SGOT (AST) or creatinine (CR)] were 1.5 times higher than the upper limit of normal value; patients with coagulation dysfunction (such as prothrombin time (PT) prolonged or shortened > 3 s, activated partial thromboplastin time (aPTT) prolonged or shortened > 10 s, platelet count (PLT) < 50 *109/L)；
5. Those with severe cardiopulmonary disease and uncontrolled epilepsy within half a year are limited to participate in the study；
6. Cervical spinal cord disease, brachial plexus nerve injury, poor compliance, psychosis, mental disorders, difficult to cooperate with；
7. Pregnancy test positive, pregnant or lactating women, recent family planning; during the trial can not take feasible contraceptive measure；
8. Surgical site peripheral nerve injury；
9. Subjects who had participated in clinical studies of other drugs, biological agents or medical devices before enrollment did not reach the primary endpoint
10. High blood pressure control is still not suitable for surgery；
11. Malignant Tumor Patients；
12. Researchers believe that there are other circumstances that are not suitable for this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-09-22 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
UCLA score | 6 months
  Efficiency of 6 months after operation=Number of subjects with excellent score + good + acceptable score / total number of subjects * 100%

SECONDARY OUTCOMES:
UCLA score | 3 months
  Efficiency of 3 months after operation=Number of subjects with excellent score + good + acceptable score / total number of subjects * 100%
constant-murley score | 3 months
  The higher the score, the better shoulder function.
ASES score | 3 months
  The higher the score, the better shoulder function.

CONTACTS AND LOCATIONS:
Locations (1):
- Full seam anchor, Hangzhou, Zhejiang, China